CLINICAL TRIAL: NCT06769347
Title: Circulating Vascular Regenerative Cell Exhaustion in Individuals Without Type 2 Diabetes Who Are of South Asian or European Origins
Acronym: ORIGINS-VRCE-2
Status: Recruiting | Type: Observational
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: Unity Health Toronto (Other); Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00083605
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases Risk
Keywords: Progenitor Cells; Cardiometabolic Risk; Ethnic Origins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Frozen and aliquoted serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- South Asian Origins: Individuals who identify as having Anglo-Indian, Bangladeshi, Bengali, Bhutanese, Goan, Gujarati, Indian, Jatt, Kashmiri, Maharashtrian, Malayali, Nepali, Pakistani, Punjabi, Sindhi, Sinhalese, Sri Lankan, Tamil, Telugu, or other South Asian origin
- European Origins: Individuals who identify as having western European, northern European, southern European, eastern European or other European origin

SUMMARY:
ORIGINS-VRCE-2 is an observational study aimed to assess how blood vessel forming stem cells from individuals without diabetes or a history of cardiovascular disease differ between individuals of South Asian and European ethnicities. The overarching objective of the study is to investigate whether differential vessel reparative stem cell populations and characteristics may underlie the elevated cardiovascular risk observed among South Asian individuals compared to individuals of European origins.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the main cause of death worldwide. Notably, individuals of South Asian (SA) origin have 3 to 5-fold increased rates of CVD compared to European individuals, which cannot be entirely explained by diet, lifestyle, or socioeconomic factors. Therefore, the mechanisms driving the increased CVD risk in SA individuals remains largely unknown.

Cardiovascular health is maintained by vascular regenerative cells, which secrete pro-vascular cytokines involved in various pro-angiogenic, arteriogenic and vasculogenic pathways. It has been shown that SA adults with type 2 diabetes or CVD show vascular regenerative cell exhaustion (VRCE), characterized by a reduced number or dysfunction of pro-vascular cells compared to European adults with type 2 diabetes or CVD. Thus, VRCE presents as a novel mechanism to explain the increased cardiovascular risk SA individuals experience. However, it is unclear whether VRCE only occurs in people with cardiometabolic diseases, or if it is a phenomenon that is also present in healthy SA individuals.

ORIGINS-VRCE-2 is an observational, two-armed, cross-sectional study that will enroll 60 healthy South Asian and 60 healthy European individuals. Vascular regenerative cells will be isolated from peripheral blood samples for enumeration and characterization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older of South Asian origin or European origin as defined by the following: i. South Asian defined as any individual who identifies as Anglo-Indian, Bangladeshi, Bengali, Bhutanese, Goan, Gujarati, Indian, Jatt, Kashmiri, Maharashtrian, Malayali, Nepali, Pakistani, Punjabi, Sindhi, Sinhalese, Sri Lankan, Tamil, Telugu, or other South Asian origins. ii. European Origin defined as any individual who identifies as from western Europe, northern Europe, southern Europe, eastern Europe or other European origins.
2. Willing and able to provide written informed consent and comply with study requirements
3. Must fulfill the following exclusion criteria:

Exclusion Criteria:

1. No previous diagnosis of type 2 diabetes
2. Any previous CV events such as:

   1. Prior myocardial infarction
   2. Coronary revascularization
   3. Coronary artery disease, peripheral artery disease, cerebrovascular disease
3. Any life-threatening disease expected to result in death within the next 2 years
4. Any malignancy not considered cured (except basal cell carcinoma of the skin). A subject is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening
5. Known severe liver disease (e.g. Non-alcoholic fatty liver disease, chronic liver disease, liver cirrhosis, etc.)
6. White blood cell count ≥ 15 x 10^9/L
7. Active infectious disease requiring antibiotic or anti-viral agents
8. Known acquired immunodeficiency syndrome such as HIV
9. On oral steroid therapy (e.g. prednisone) or other immunosuppressive agents (e.g. methotrexate)
10. Treated autoimmune disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from primary care and cardiology outpatient clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The differences in the frequency / absolute number of circulating ALDHhi primitive progenitor cells co-expressing CD133 between individuals of South Asian origins and European origins | Baseline

SECONDARY OUTCOMES:
The differences in the frequency / absolute number of circulating ALDHhiSSCmid precursor cells with monocytes/macrophage phenotype between individuals of South Asian origins and European origin | Baseline

OTHER OUTCOMES:
Difference in the amount of intracellular reactive oxygen species (ROS) production in ALDHhi progenitor cell subsets in individuals of South Asian origins and European origins | Baseline
Difference in the levels of inflammatory and oxidative stress biomarkers in individuals of South Asian origins and European origins | Baseline

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Markham HealthPlex Medical Centre, Markham, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Marlee Medical Centre, North York, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario
  - Langstaff Medical Centre, Woodbridge, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Capoccia BJ, Robson DL, Levac KD, Maxwell DJ, Hohm SA, Neelamkavil MJ, Bell GI, Xenocostas A, Link DC, Piwnica-Worms D, Nolta JA, Hess DA. Revascularization of ischemic limbs after transplantation of human bone marrow cells with high aldehyde dehydrogenase activity. Blood. 2009 May 21;113(21):5340-51. doi: 10.1182/blood-2008-04-154567. Epub 2009 Mar 26. PMID 19324906
- [Background] Putman DM, Liu KY, Broughton HC, Bell GI, Hess DA. Umbilical cord blood-derived aldehyde dehydrogenase-expressing progenitor cells promote recovery from acute ischemic injury. Stem Cells. 2012 Oct;30(10):2248-60. doi: 10.1002/stem.1206. PMID 22899443
- [Background] Krishnaraj A, Bakbak E, Teoh H, Pan Y, Firoz IN, Pandey AK, Terenzi DC, Verma R, Bari B, Bakbak AI, Kunjummar SP, Yanagawa B, Connelly KA, Mazer CD, Rotstein OD, Quan A, Bhatt DL, McGuire DK, Hess DA, Verma S. Vascular Regenerative Cell Deficiencies in South Asian Adults. J Am Coll Cardiol. 2024 Feb 20;83(7):755-769. doi: 10.1016/j.jacc.2023.12.012. PMID 38355246
- [Background] Bakbak E, Verma S, Krishnaraj A, Quan A, Wang CH, Pan Y, Puar P, Mason T, Verma R, Terenzi DC, Rotstein OD, Yan AT, Connelly KA, Teoh H, Mazer CD, Hess DA. Empagliflozin improves circulating vascular regenerative cell content in people without diabetes with risk factors for adverse cardiac remodeling. Am J Physiol Heart Circ Physiol. 2023 Nov 1;325(5):H1210-H1222. doi: 10.1152/ajpheart.00141.2023. Epub 2023 Sep 29. PMID 37773589
- [Background] Hess DA, Trac JZ, Glazer SA, Terenzi DC, Quan A, Teoh H, Al-Omran M, Bhatt DL, Mazer CD, Rotstein OD, Verma S. Vascular Risk Reduction in Obesity through Reduced Granulocyte Burden and Improved Angiogenic Monocyte Content following Bariatric Surgery. Cell Rep Med. 2020 May 19;1(2):100018. doi: 10.1016/j.xcrm.2020.100018. eCollection 2020 May 19. PMID 33205058
- [Background] Terenzi DC, Trac JZ, Teoh H, Gerstein HC, Bhatt DL, Al-Omran M, Verma S, Hess DA. Vascular Regenerative Cell Exhaustion in Diabetes: Translational Opportunities to Mitigate Cardiometabolic Risk. Trends Mol Med. 2019 Jul;25(7):640-655. doi: 10.1016/j.molmed.2019.03.006. Epub 2019 Apr 30. PMID 31053416
- [Background] Terenzi DC, Bakbak E, Trac JZ, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Isolation and characterization of circulating pro-vascular progenitor cell subsets from human whole blood samples. STAR Protoc. 2021 Feb 1;2(1):100311. doi: 10.1016/j.xpro.2021.100311. eCollection 2021 Mar 19. PMID 33554145
- [Background] Patel AP, Wang M, Kartoun U, Ng K, Khera AV. Quantifying and Understanding the Higher Risk of Atherosclerotic Cardiovascular Disease Among South Asian Individuals: Results From the UK Biobank Prospective Cohort Study. Circulation. 2021 Aug 10;144(6):410-422. doi: 10.1161/CIRCULATIONAHA.120.052430. Epub 2021 Jul 12. PMID 34247495
- [Background] Volgman AS, Palaniappan LS, Aggarwal NT, Gupta M, Khandelwal A, Krishnan AV, Lichtman JH, Mehta LS, Patel HN, Shah KS, Shah SH, Watson KE; American Heart Association Council on Epidemiology and Prevention; Cardiovascular Disease and Stroke in Women and Special Populations Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Atherosclerotic Cardiovascular Disease in South Asians in the United States: Epidemiology, Risk Factors, and Treatments: A Scientific Statement From the American Heart Association. Circulation. 2018 Jul 3;138(1):e1-e34. doi: 10.1161/CIR.0000000000000580. Epub 2018 May 24. PMID 29794080
- [Background] Gupta M, Singh N, Verma S. South Asians and cardiovascular risk: what clinicians should know. Circulation. 2006 Jun 27;113(25):e924-9. doi: 10.1161/CIRCULATIONAHA.105.583815. No abstract available. PMID 16801466
- [Background] GBD 2021 Diabetes Collaborators. Global, regional, and national burden of diabetes from 1990 to 2021, with projections of prevalence to 2050: a systematic analysis for the Global Burden of Disease Study 2021. Lancet. 2023 Jul 15;402(10397):203-234. doi: 10.1016/S0140-6736(23)01301-6. Epub 2023 Jun 22. PMID 37356446
- [Background] Vaduganathan M, Mensah GA, Turco JV, Fuster V, Roth GA. The Global Burden of Cardiovascular Diseases and Risk: A Compass for Future Health. J Am Coll Cardiol. 2022 Dec 20;80(25):2361-2371. doi: 10.1016/j.jacc.2022.11.005. Epub 2022 Nov 9. No abstract available. PMID 36368511